## Janssen Research & Development

### **Statistical Analysis Plan**

## Continued access to etravirine in treatment experienced HIV-1 infected subjects.

#### Protocol TMC125-TiDP35-C239; Phase N/A

TMC125 Intelence®/(Etravirine)

Status: Approved

**Date:** 20 January 2021

Prepared by: Janssen Research & Development, LLC

**Document No.:** EDMS-RIM-305084, 3.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

# **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

Approved, Date: 20 January 2021

# **TABLE OF CONTENTS**

| TAB | BLE OF CONTENTS | <mark>2</mark> |
|---|---|---|
| AME | ENDMENT HISTORY | 3 |
| ABB | BREVIATIONS | 3 |
| 1. | INTRODUCTION | 4 |
| 1.1. | Trial Objectives | |
| 1.2. | Trial Design | 4 |
| 1.3. | Statistical Hypotheses for Trial Objectives | 6 |
| 1.4. | Sample Size Justification | 6 |
| 1.5. | Randomization and Blinding | 6 |
| 2. | GENERAL ANALYSIS DEFINITIONS | 6 |
| 2.1. | Analysis Sets | |
| 2.1.1 | | |
| 2.2. | Study Day and Relative Day | |
| 2.3. | Baseline and Endpoint | |
| 2.4. | General Analysis Rules | |
| 3. | INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW | <b>7</b> |
| 4. | COVID RELATED DEVIATIONS | <mark>7</mark> |
| 5. | SUBJECT INFORMATION | 7 |
| 5.1. | Demographics and Baseline Characteristics | |
| 5.2. | Disposition Information | |
| 5.3. | Treatment Compliance | 8 |
| 5.4. | Extent of Experies | _ |
| | Extent of Exposure | 8 |
| 5.5. | Protocol Deviations | 8 |
| 5.6. | Protocol Deviations | 8<br>8 |
| 5.6.<br>Will | Protocol Deviations Prior and Concomitant Medications be summarized by CMDECODE antiretroviral category | 8<br>88 |
| 5.6.<br>Will | Protocol Deviations | 8<br>88 |
| 5.5.<br>5.6.<br>Will<br>5.7. | Protocol Deviations Prior and Concomitant Medications be summarized by CMDECODE antiretroviral category | 8<br>8<br>8 |
| 5.6.<br>Will<br>5.7. | Protocol Deviations Prior and Concomitant Medications be summarized by CMDECODE antiretroviral category Medical history | 8<br>8<br>8 |
| 5.6.<br>Will<br>5.7.<br><b>6.</b><br><b>7.</b> | Protocol Deviations Prior and Concomitant Medications be summarized by CMDECODE antiretroviral category Medical history EFFICACY SAFETY Adverse Events | 8<br>8<br>8 |
| 5.6.<br>Will<br>5.7.<br><b>6.</b> | Protocol Deviations Prior and Concomitant Medications be summarized by CMDECODE antiretroviral category Medical history EFFICACY SAFETY | 8<br>8<br>8 |

### **AMENDMENT HISTORY**

Not applicable

#### **ABBREVIATIONS**

AE adverse event

ATC anatomic and therapeutic Class

BMI body mass index body surface area BSA confidence interval CI CRF case report form Clinical Study Report **CSR** coefficient of variation CVDMC Data Monitoring Committee **DPS** Data Presentation Specifications

ECG electrocardiogram

eCRF electronic case report form

FAS full analysis set

FDA Food and Drug Administration

ICH International Conference on Harmonization

IQ interquartile

MedDRA Medical Dictionary for Regulatory Activities

PD pharmacodynamic
PK pharmacokinetic(s)
SAE serious adverse event
SAP Statistical Analysis Plan
SD standard deviation

SMQs standardised MedDRA queries
TEAE treatment-emergent adverse event
WHO World Health Organization

WHO-DD World Health Organization Drug Dictionary

ITT Intention-to-Treat

### 1. INTRODUCTION

This is a continued access trial for subjects who have completed treatment in a clinical trial with ETR sponsored by or in collaboration with Janssen Research & Development, and who continue to benefit from the use of ETR.

This statistical analysis plan (SAP) for the TMC125-TiDP35-C239 describes the statistical analysis for subject information and safety data.

## 1.1. Trial Objectives

The primary objective of the trial is to continue to provide ETR to subjects who previously received ETR in a clinical trial and continue to benefit from the use of ETR, in countries where ETR is not commercially available for the subject's indication, is not reimbursed, and cannot be accessed through another source (e.g. access program or government program), or where the subject is not eligible for ongoing trials/programs with ETR.

# 1.2. Trial Design

At the baseline visit, inclusion/exclusion criteria will be checked to confirm eligibility. Once eligibility criteria are met, subjects will either continue on the ETR dose they have received in the previous ETR trial or on an adjusted dose if deemed necessary by the investigator. For pediatric subjects, ETR dose adjustment will be based on weight using the dosing guidelines provided.

Assessment visits are recommended according to local generally accepted standard of care, but not less frequent than every three and six months for pediatric and adult subjects respectively. Adverse events leading to discontinuation or treatment interruption, adverse events at least possibly related to treatment with ETR, serious adverse events, and pregnancies will be recorded at each visit. In addition to the assessments described in the flowchart, additional assessments not included in this protocol can be done locally at the investigator's discretion as per local standard of care.

Treatment will be continued until one of the following criteria is met: the investigator determines that the subject no longer benefits from ETR treatment (e.g., based on viral load); treatment limiting toxicity; loss to follow-up; patient withdrawal of consent; pregnancy; termination of the program by the Sponsor; ETR becomes commercially available for the subject's indication, is reimbursed, or can be accessed through another source (e.g. access program, government program) in the region the subject is living in, whichever occurs first. A diagram of the study design is provided below in Figure 1.

Figure 1: Schematic Overview of the Study

| Type of Visit | Baseline | | Treatment p | period | Follow-up |
|---|---|---|---|---|---|
| Time of Visit | Day 1 | Every 3<br>months<br>for<br>pediatric | Every 6<br>months for<br>adult<br>subjects | Final /<br>withdrawal<br>visit <sup>c</sup> | 4 weeks<br>after<br>withdrawal |
| Informed Consent/Assent <sup>g</sup> | X | | | | |
| Demographic data <sup>d</sup> | X | | | | |
| Height <sup>h</sup> , Tanner staging <sup>h</sup> | X | | | X | |
| Weight | X | X | X | | |
| Urine pregnancy test, if applicable <sup>e</sup> | X | X | X | X | |
| Inclusion/exclusion criteria | X | | | | |
| Dispensation of investigational medication | X | X | X | | |
| Drug accountability | | X | X | X | |
| Collection of the following AEs <sup>f</sup> : - AEs considered to be at least possibly related to ETR; | X | X | X | X | X |
| - AEs leading to discontinuations or treatment interruption; | | | | | |

- a Subject will rollover from another trial. Baseline visit will coincide with the last visit of the previous trial. Assessments and results from the last visit of the previous trial will be used for the Baseline Visit of this trial.
- b Only for subjects who drop out of the study due to the occurrence of a (S)AE.
- c Any AE event ongoing at the end of treatment should be followed up until satisfactory clinical resolution or stabilization at the investigator's discretion, according to the local standard of care.
- d Including Subject ID from feeder trial.
- e Urine pregnancy test for females of childbearing potential only.
- f Other AEs will only be collected if required per local regulations.
- g Informed assent only applicable to pediatric subjects.
- h Only applicable to pediatric subjects.

### 1.3. Statistical Hypotheses for Trial Objectives

N/A

## 1.4. Sample Size Justification

No formal sample size calculation has been performed. The trial is not set up to show a specific statistical hypothesis but to provide ETR to subjects who previously received ETR in a clinical trial sponsored by Janssen Research & Development, and continue to benefit from the use of ETR, in countries where ETR is not commercially available to subjects, is not reimbursed, and is not accessible through another source (e.g. access program or government program), or where the subject is not eligible for ongoing trials/programs with ETR. Data from this trial may be included in Safety Updates.

### 1.5. Randomization and Blinding

Since this is an open-label trial, blinding procedures are not applicable.

#### 2. GENERAL ANALYSIS DEFINITIONS

# 2.1. Analysis Sets

Intent-to-treat (ITT) population: the set of all subjects who have taken at least 1 dose of ETR, regardless of their compliance with the protocol and adherence to the dosing regimen.

## 2.1.1. Safety Analysis Set

All safety results will be presented for the ITT population.

# 2.2. Study Day and Relative Day

Study Day 1 or Day 1 refers to the start of the first study agent administration. All safety assessments at all visits will be assigned a day relative to this date.

Study day or relative day for a visit is defined as:

- Visit date (date of Study Day 1) +1, if visit date is ≥date of Day 1
- Visit date Date of Day 1, if visit date <date of Day 1

There is no 'Day 0'

# 2.3. Baseline and Endpoint

Baseline is defined as the last observation prior to the start of the first study agent administrations.

### 2.4. General Analysis Rules

• Data of adult and pediatric subjects will be analyzed separately. For the statistical analysis of TMC125-C239, a pediatric and adult subject will be defined as a subject who entered the previous trial at age < 18 and ≥ 18 years old respectively. Subjects who turn 18 while in the

previous trial or in TMC125-C239 will be considered as pediatric subjects for the statistical analysis.

- Continuous data will be summarized by descriptive statistics, including number of subjects (N), mean, standard deviation (SD), median, and range (minimum; maximum).
- The minimum and maximum will be presented to the same number of decimal places as the original data. The mean, median and 95% CI will be rounded to one additional decimal place than the original data, while SD will be approximated to two additional decimal places.
- If a count is 0, the percentage (0%) should not be displayed. The 0 count will be displayed, but the corresponding percentage should be omitted.
- The percentages (%) in tables will be presented to 1 decimal place unless the sample sizes for the percentages are small enough to warrant presenting as integers.

### 3. INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW

There is no interim analysis planned for this study.

### 4. COVID RELATED DEVIATIONS

All COVID related deviations will be tabulated and listed.

#### 5. SUBJECT INFORMATION

# 5.1. Demographics and Baseline Characteristics

Table 01 presents a list of the demographic variables that will be summarized by pediatric and adult subjects separately as well as all combined for ITT analysis set.

**Table 01: Demographic Variables** 

| Continuous Variables | Summary Type |
|-----------------------|------------------------------|
| Age (years) | Descriptive statistics (N, |
| Height (cm) | mean, standard deviation |
| Weight (kg) | [SD], median and range |
| | [minimum and maximum]) |
| Categorical Variables | |
| Sex (male, female) | Frequency distribution with |
| | the number and percentage of |
| | subjects in each category. |

The demographics and baseline characteristics will be listed for all subjects.

### 5.2. Disposition Information

The number of subjects in the following disposition categories will be summarized:

- Subject didn't fulfill all inclusion/exclusion criteria (screen failures)
- AE/HIV-related event/Cutaneous event/Rash (including death, abnormal lab values, current illnesses)

7

- Lost to follow-up
- Withdrew consent/assent
- Non-compliant
- Ineligible to continue the trial
- Investigator no longer thinks subject benefits from the ETR treatment
- Sponsor's decision
- Switch to commercially available medication
- Other

## 5.3. Treatment Compliance

Not applicable for this study

### 5.4. Extent of Exposure

Not applicable for this study

#### 5.5. Protocol Deviations

If captured, major protocol deviations will be defined. A listing of subjects with a major protocol deviation will be provided.

#### 5.6. Prior and Concomitant Medications

Will be summarized by CMDECODE antiretroviral category

### 5.7. Medical history

Not applicable

# 6. EFFICACY

N/A

#### 7. SAFETY

All safety analyses will be based on the safety analysis set.

Safety data of adult and pediatric subjects will be analyzed separately as well as overall.

For all continuous safety variables, descriptive statistics will include the N, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized using frequency counts and percentages.

#### 7.1. Adverse Events

The verbatim terms used in the CRF by investigators to identify adverse events will be coded using the available version of the Medical Dictionary for Regulatory Activities (MedDRA version 23.0). Treatment-emergent adverse events are adverse events with onset during the treatment phase or

that are a consequence of a pre-existing condition that has worsened since baseline. If the event occurs on the day of the initial administration of study agent, and either event time or time of administration are missing, then the event will be assumed to be treatment emergent. If the event date is recorded as partial or completely missing, then the event will be considered treatment emergent unless it is known to be prior to the first administration of study agent based on partial onset date or resolution date. All reported adverse events will be included in the analysis. For each adverse event, the number and percentage of subjects who experience at least 1 occurrence of the given event will be summarized by treatment.

Summary tables will be provided by pediatric and adult subjects separately as well as overall for:

- Mortality
- Serious AEs (SAEs)
- AEs leading to discontinuation of treatment
- AEs possibly related to ETR
- All AEs

From the collected (S)AE data in TMC125-C239, the following events will be summarized:

## Skin events

Skin events of interest will be assigned to categories from the following list:

- '(Serious) Rash Cases': a predefined list of selected PTs used for the post-marketing safety monitoring, is used to identify (serious) cases of Rash.

Acrodynia Rash generalised Drug eruption Rash macular Erythema ab igne Rash maculo-papular Erythema Rash maculovesicular Erythema elevatum diutinum Rash morbilliform Erythema toxicum neonatorum Rash neonatal Fixed eruption Rash papular Generalised erythema Rash pruritic Lupus miliaris disseminates faciei Rash pustular Mucocutaneous rash Rash rubelliform Necrolytic migratory erythema Rash scarlatiniform Rash Red man syndrome Rash vesicular Rash erythematous

- '(Severe) Cutaneous Reactions': the MedDRA SMQ (Severe) Cutaneous Adverse Reactions [Broad scope SMQ code: 20000020], which includes Stevens-Johnson Syndrome, is used
  - to identify cases.
- 'Angioedema': the MedDRA SMQ Angioedema (SMQ, broad) is used to identify cases.

- Cardiac
- Hepatobilliary

#### Hepatic events

Hepatic events of interest (or 'Hepatotoxicity') will be assigned to the subcategories from the following list, with relevant SMQs to identify cases:

- "Cholestasis and jaundice": Cholestasis and jaundice of hepatic origin, broad (SMQ code: 20000009),
- "Hepatic Failure, fibrosis and cirrhosis and other": Hepatic failure fibrosis and cirrhosis and other liver damage-related conditions, broad (SMQ code: 20000013),
- "Hepatitis non-infectious": Hepatitis non-infectious, broad (SMQ code: 20000010),
- "Liver related investigations, signs and symptoms": Liver related investigations signs and symptoms, broad (SMQ code: 20000008).
  - Neuropsychiatric

In addition to the summary tables, listings will be provided for subjects who:

- Mortality
- Had SAEs
- Had AEs leading to discontinuation of treatment

# 7.2. Clinical Laboratory Tests and Vital Signs Findings

#### Missing baseline values:

The only reference time point for the weight analysis will be baseline. If there is no baseline value available, no changes will be calculated. Observed and change from baseline in weight by visit will be summarized by pediatric and adult subjects separately. Table 2 and Table 3 show the definition of windows used for the weight analysis for pediatric and adult, respectively.

Table 2: Definition of windows for weight (pediatric subjects)

| Phase | Visit | Target day | Analysis time point | Time interval (days) |
|---|---|---|---|---|
| Baseline | 1 | 1 | Baseline | <=1 |
| Treatment | 2 | 90 | Month 3 | 2 to 135 |
| | 3 | 180 | Month 6 | 136 to 225 |
| | 4+ | XX*30 | Month XX | [XX*30 days – 44 to XX*30 days + 45] |

Table 3: Definition of windows for weight (adult subjects)

| Phase | Visit | Target day | Analysis time point | Time interval (days) |
|---|---|---|---|---|
| Baseline | 1 | 1 | Baseline | <=1 |
| Treatment | 2 | 180 | Month 6 | 2 to 270 |
| | 3 | 360 | Month 12 | 271 to 450 |
| | 4+ | XX*30 | Month XX | [XX*30 days – 89 to XX*30 days + 90] |

If two (or more) measurements fall within the same time interval, the measurement closest to the target day (in case of equal distances, latest measurement takes precedence) is used for the analysis displays and graphics in order to have only one measurement per subject per analysis time point. However, all data are presented in the listings.

The number of days in the treatment is defined as:

relday = visit day – reference day+1 for visits on or after the reference

relday = visit day – reference day for visits before the reference where the reference day equals the actual start date of intake of ETR.

### 7.3. Overview of statistical output

| COVID related deviations | |
|---|---|
| TCOV01 | COVID-related deviations: Tabulation |
| LCOV01 | COVID-related deviations: Listing |
| Demographics | |
| TDEM01 | Demographics and baseline characteristics |
| LDEM01 | Listing of demographics and baseline characteristics |
| Prior and Concomitant Medications | |
| TSICM01 | Prior ARV Therapies; Individual ARVs |
| TSICM02a | Initial OBR Therapies Individual ARVs |
| TSICM02b | Initial OBR Therapies Combinations of ARVs |
| Disposition | |
| TDIS01 | Disposition |

11

| LDIS01 | Listing of disposition |
|---|---|
| Safety | |
| TSFAE01 | Adverse Events: Summary Table |
| TSFAE02 | Adverse Events: Tabulation of All Events by System Organ Class and Preferred Term |
| TSFAE03 | Frequency (%) of Serious Adverse Events |
| TSFAE04 | Frequency (%) of Grade 3-4 Adverse Events (Regardless of Causality) |
| TSFAE05 | Frequency (%) of Adverse Events at Least Possibly Related to Etravirine |
| TSFAE06 | Frequency (%) of Adverse Events Leading to Permanent Stop of Study Medication |
| TSFAE07 | Adverse Events of Interest by Event of Interest Group |
| LSFAE01 | Adverse Events: Summary Listing of All Events |
| LSFAE02 | Adverse Events: All Events with Grade 3 to 4 Toxicity |
| LSFAE03 | Adverse Events: All Serious Events |
| LSFAE04 | Adverse Events: All Events at Least Possibly Related to Study Medication |
| LSFAE05 | Adverse Events of Interest: Summary Listing of All Events of Interest |
| LSFAE06 | Adverse Events: All Events Leading to Permanent Stop of Study Medication |
| TSFVIT01a | Observed and Change from Baseline in Weight by visit (pediatric) |
| TSFVIT01b | Observed and Change from Baseline in Weight by visit (adult) |
| TSLWT01a | Listing: Weight (pediatric) |
| TSLWT01b | Listing: Weight (adult) |